CLINICAL TRIAL: NCT00242047
Title: Randomized, Controlled Trial Comparing Efficacy of Percutaneous and Intradermal Vaccination With Japanese (Tokyo) 172 BCG in the Prevention of Tuberculosis In Infants Vaccinated at Birth
Brief Title: Randomized Controlled Trial of Percutaneous and Intradermal BCG Vaccination.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cape Town (Other)
Collaborators: Aeras (Other); Japan BCG Laboratory 4-2-6 Kohinata,Tokyo 112-0006, Japan. (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UCT REC 271/2000
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2005-10-19 (Estimated); Status verified 2004-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis.; Children.; Vaccine.; BCG.
MeSH Terms: conditions — Tuberculosis

INTERVENTIONS:
Biological: Japanese (Tokyo) 172 Bacille Calmette Guerin (BCG).

SUMMARY:
An open label, randomized, controlled, equivalency trial to compare the efficacy of the percutaneous route of administration with the intradermal route of administration of Japanese (Tokyo) 172 BCG, in the prevention of tuberculosis during the first two years of life.

DETAILED DESCRIPTION:
This is an open label, randomized, controlled, equivalency trial to compare the efficacy of the percutaneous route of administration with the intradermal route of administration of Japanese (Tokyo) 172 BCG, obtained from the BCG laboratory in Tokyo, Japan, in the prevention of tuberculosis, with bacteriological or histological confirmation, or meeting strict clinical criteria, during the first two years of life. The comparison of the two methods is necessary because the intradermal method is almost universally preferred, without direct evidence from a clinical trial. The intradermal method provides for more accurate dosing and produces a higher rate of tuberculin skin test conversion, but neither of these factors has been shown to correlate with efficacy of BCG vaccination. The percutaneous method is much simpler and, if shown to be equally effective, could become a preferred method. The Japanese strain was chosen because it is the one commercially available strain produced for both intradermal and percutaneous administration, and because a seed lot from this strain was previously used to produce BCG for the South African BCG vaccination program.

ELIGIBILITY:
Inclusion Criteria:

1. The child must be eligible to receive routine BCG vaccination.
2. The child must be born at one of the five hospitals taking part in the study and be a resident in the study area.
3. The mother must have had an opportunity to become informed about the study, either through pre-natal classes and a follow-up visit or, if time and the situation permits, after the mother presents at the hospital or birthing facility and before or after the child is born.
4. After being informed about the study, the mother gives consent for the infant to be enrolled and signs a consent form.

Exclusion Criteria:

1. The mother fails to give informed consent.
2. The child has a medical condition which contraindicates vaccination during the first 24 hours of life (e.g., birth weight below 2,500 grams).
3. The infant is hospitalized outside of the study area before vaccination has been given (e.g. transferred to a hospital in Cape Town because of respiratory distress).

Ages: 0 Years to 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12000
Dates: Start 2001-03; Study Completion 2006-08

PRIMARY OUTCOMES:
Prevention of tuberculosis with bacteriological or histological confirmation, or meeting strict clinical criteria,in the first 2 years of life.

SECONDARY OUTCOMES:
Comparison of Rate of Adverse Events.
Comparison of Mortality Rates.
Microbiological diagnosis of tuberculosis in a primary care setting.
Rating of diagnostic scoring systems.
Case definition of tuberculosis.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hussey, FCCH, Principal Investigator — South African Tuberculosis Vaccine Initiative; Larry Geiter, PhD, Principal Investigator — Aeras
Locations (1):
- South African Tuberculosis Vaccine Initiative, Institute of Infectious Disease and Molecular Medicine, University of Cape Town., Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Hawkridge A, Hatherill M, Little F, Goetz MA, Barker L, Mahomed H, Sadoff J, Hanekom W, Geiter L, Hussey G; South African BCG trial team. Efficacy of percutaneous versus intradermal BCG in the prevention of tuberculosis in South African infants: randomised trial. BMJ. 2008 Nov 13;337:a2052. doi: 10.1136/bmj.a2052. PMID 19008268
- See also: SATVI website — http://www.satvi.uct.ac.za/